CLINICAL TRIAL: NCT02914340
Title: REACH (Research to Assess SVS Safety and Effectiveness for the Treatment of Severe EmphysemA in China) SVS Control Patient Cross-Over Study
Brief Title: REACH SVS Control Patient Cross-Over Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR-04524
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): The treatment algorithm is complete occlusion of one lobe of the lung by using valves to occlude all segments of the lobe. The lobe will be selected based on imaging with high resolution computed tomography (HRCT). The lobe to be treated will have severe heterogeneous emphysema based on visual exam. The selected lobe will also have an intact fissure separation with the ipsilateral lobe. An intact fissure will be estimated visually to be ≥ 90% complete after viewing the HRCT in 3 dimensions. If more than one lobe meets criteria, the investigator will determine a primary lobe to treat based on fissure completeness, heterogeneity, disease severity, and the anatomy of the airways that will be treated.
  Interventions: Device: Spiration Valve System

INTERVENTIONS:
Device: Spiration Valve System

SUMMARY:
This is a multicenter, prospective study designed to evaluate performance of the SVS in the REACH SVS control patients. The study is expected to enroll up to 20 patients at up to 12 sites with up to 6 patients per site.

ELIGIBILITY:
Inclusion Criteria:

* Patient was enrolled in the REACH SVS Study control group and has completed their participation in the Study including the 12 month follow-up visit.
* Patient has received standard-of-care medical management and it has been stable for 6 weeks.
* Patient is willing to participate in a study, complete the required follow-up visits, and maintain consistent nutrition and exercise habits during the study period.

Exclusion Criteria:

* Patient is classified as ASA Class greater than P4 including presence of co-morbidity that could significantly increase the risk of a bronchoscopy procedure.
* Patient participated in a study of an investigational drug or device within the past 30 days prior to participation in this study.
* Patient has demonstrated unwillingness or inability to complete baseline data collection procedures.
* Patient has co-existing major medical disease that will limit evaluation, participation, or follow-up in the study.
* Patient is unable to provide informed consent.
* Patient is not an appropriate candidate for or is unable to tolerate, flexible bronchoscopy procedures.
* Patient has history of 4 or more hospitalizations for COPD exacerbation or respiratory infections in the past year and none have occurred in the prior 3 months.
* Patient has evidence of systemic disease or neoplasia expected to compromise survival during the 3-month study period
* Patient has demonstrated unwillingness or inability to complete screening or baseline data collection procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume at 1 second | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided